CLINICAL TRIAL: NCT04158206
Title: Explored Maternal Voice on Alleviating Pain in Premature Undergoing Heel Lance Procedure and Enhancing Mother-Infant Bonding
Brief Title: Maternal Voice on Alleviating Pain in Premature Undergoing Heel Lance Procedure and Enhancing Mother-Infant Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1902160001
Record Dates: First submitted 2019-10-18; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Infant, Extremely Premature; Voice; Pain; Bonding
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal voice (Experimental): The mother's voice recordings are compiled for 13 minutes. When the premature infants undergoing heel lance procedure, the experimental group were explored maternal voice, which start from 3 minutes before the procedure, once a day and for three consecutive days.And then recorded the process by the camera, uploaded to YouTube within 24 hours and sent to their mother.
  Interventions: Other: Maternal voice
- control group (No Intervention): When the premature infants undergoing heel lance procedure, the control group were under routine care.And then recorded the process by the camera for three consecutive days, uploaded to YouTube within 24 hours and sent to their mother.

INTERVENTIONS:
Other: Maternal voice — Recording in the intensive care unit quiet and separate consultation room. For infants in the 'maternal voice group,' mothers were asked to tape what the mother wants to say to their babies and read of a child book from the independent publish, 'Xiao Qi's yellow persimmon' which talk about the mother who has a premature infants how to take caring of their baby. After reviewing the quality of the recording, the mother's voice recordings are compiled for 13 minutes with Sound Organizer. 2 , and the volume of the sound standard according to the American Academy of Pediatrics guidelines is 60 decibels in the incubator.
  Arms: Maternal voice

SUMMARY:
A total of 64 preterm infants born before 37 weeks of gestation and their mothers were randomly assigned to the experimental and control groups. The intervention used in the experimental group involved an audio recording with repeated clips of the mother reading a children's book, edited to a duration of 13 minutes. The research commenced on the fourth day after the birth of the research subjects, in which the maternal voice recording was played to infants during heel lance procedure once a day for 3 consecutive days. The infants in the control group received general routine care during heel lance procedure. Physiological indicators, including heart rate, respiratory rate, oxygen saturation, and pain response assessed using the Neonatal Infants Pain Scale (NIPS), were recorded 3 minutes before, during, and at the first and 10th minute after heel lance procedure. From the fourth to the sixth day after birth, video recordings of the research process were made and sent to the mother for viewing. On the seventh day after birth, the effectiveness of mother-infant bonding was evaluated using the Mother-Infant Bonding Inventory (MIBI).

DETAILED DESCRIPTION:
This study is a quantitative study, using Experimental Research Design, using G*Power 3.1 to estimate the number of samples, the sample size is 62. There aren't rule out the possibility of congenital hearing loss. According to the literature, the prevalence of deafness in premature or low-weight newborns is about 1-2%. Therefore, the number of samples will increase by 2 according to the prevalence of deafness. After the completion of the case, the hearing screening of the subjects will be continuously tracked to avoid the final loss of samples. Therefore, the total number of cases is 64. In this study, the allocation concealment principle was applied. Before the distribution, the main caregivers and researchers did not know the distribution rules and the distribution results. The sampling method of randomized control trial stratified block randomization was adopted. According to the past clinical birth rate, the number of weeks of pregnancy was less than 31+6 weeks. The proportion of newborns born from 32 weeks to 36+6 weeks of gestational weeks is about 1:2, respectively. Finally, the experimental group and the control group were randomly assigned in this way. There are 20 infants in less than 31+6 weeks group, 44 infants in more than 31+6 weeks group.

The process of receiving the case was the evening of the 4th day after the birth of the study subjects. The premature infants of the experimental group began to listen the maternal voice 3 minutes before the heel lance procedure until the end of the blood collection for 13 minutes, Heart rate (HR), respiratory rate (RR), oxygen saturation (%, OSPR), and pain which evaluated by Neonatal Infants Pain Scale (NIPS) were recorded 3 minutes before, during,and at the first and 10th minutes after heel lance procedure. The monitoring was continued for 3 days.

The study was conducted for three consecutive days from the fourth day after the birth of the subject. The three-day experimental group and the control group were recorded by the camera, uploaded to YouTube within 24 hours after recording, and the film was used for three consecutive days using a private link. Confirm that the mother has watched this video.and please ask the mother to fill out the mother-infant bonding questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1.Babies born alive before 37 weeks of pregnancy 2.Infant was singlet 3.Infants who were required to receive heel lance procedure every 8 hours after physicians' diagnoses 4.Infants' primary caregivers who could read Chinese that agreed to participate in this study and sign written consent forms

Exclusion Criteria:

* 1.Infants with congenital anomaly, congenital or postnatal sepsis, or brain injury 2.Infants' mother smoked, drunk or illegally used drugs while she was pregnant

Ages: 4 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from Baseline Heart rate at 3 minutes before, during, and at the first and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP60 Dräger Julian physiological index monitor, including monitoring Heart Rate (HR), recorded every 12 seconds.
Respiratory rate | Change from Baseline Respiratory rate at 3 minutes before, during, and at the first and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP60 Dräger Julian physiological index monitor, including monitoring Respiratory Rate (RR), recorded every 12 seconds.
Oxygen Saturation | Change from Baseline Oxygen Saturation at 3 minutes before, during, and at the first and 10th minute after heel lance procedure
  Using the German-made PHILIPS IntelliVue MP60 Dräger Julian physiological index monitor, including monitoring Saturation of Peripheral Oxygen (SPO2), recorded every 12 seconds.
Respond of Pain | Change from Baseline Pain at 3 minutes before, during, and at the first and 10th minute after heel lance procedure
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.

SECONDARY OUTCOMES:
Mother-Infant Bonding Inventory (MIBI) | On the 7th day birth
  This scale consists of three aspects, namely " proximity ", " commitment ", "confidence of reciprocity", each with 7 questions, 6 questions, 6 questions, and a total of 19 questions. The scales are all Likert-style six-point scales. The options are "very disagree", "disagree", "a little disagree", "a little agree", "agree" to "very agree", in order 1, 2, 3, 4, 5, 6 points. The score range is 19-114 points, the higher scores, the better the bonding.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Provenzi L, Broso S, Montirosso R. Do mothers sound good? A systematic review of the effects of maternal voice exposure on preterm infants' development. Neurosci Biobehav Rev. 2018 May;88:42-50. doi: 10.1016/j.neubiorev.2018.03.009. Epub 2018 Mar 10. PMID 29535067
- [Background] Chirico G, Cabano R, Villa G, Bigogno A, Ardesi M, Dioni E. Randomised study showed that recorded maternal voices reduced pain in preterm infants undergoing heel lance procedures in a neonatal intensive care unit. Acta Paediatr. 2017 Oct;106(10):1564-1568. doi: 10.1111/apa.13944. Epub 2017 Jul 5. PMID 28580602
- [Background] Filippa M, Panza C, Ferrari F, Frassoldati R, Kuhn P, Balduzzi S, D'Amico R. Systematic review of maternal voice interventions demonstrates increased stability in preterm infants. Acta Paediatr. 2017 Aug;106(8):1220-1229. doi: 10.1111/apa.13832. Epub 2017 Apr 19. PMID 28378337
- [Derived] Yu WC, Chiang MC, Lin KC, Chang CC, Lin KH, Chen CW. Effects of maternal voice on pain and mother-Infant bonding in premature infants in Taiwan: A randomized controlled trial. J Pediatr Nurs. 2022 Mar-Apr;63:e136-e142. doi: 10.1016/j.pedn.2021.09.022. Epub 2021 Sep 30. PMID 34602338